CLINICAL TRIAL: NCT06257966
Title: A Phase 3, Multi-center, Open-label, Randomized Study to Evaluate the Efficacy and Safety of JY09 Versus Dulaglutide in Patients With T2DM Inadequately Controlled by Metformin
Brief Title: A Phase 3 Study to Evaluate the Efficacy of JY09 Compared With Dulaglutide in Combination Therapy Diabetes Mellitus Type 2 Patients With Metformin
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Dongfang Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFBT-JY09-DM-302
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Type2 Diabetes Mellitus
Keywords: T2DM
MeSH Terms: interventions — dulaglutide; Metformin

STUDY DESIGN:
Intervention Model Description: Randomized in a 1:1:1 ratio to the 1.2 mg JY09 injection group (n=200 cases), the 2.4 mg JY09 injection group (n=200 cases), and the dulaglutide injection group (n=200 cases).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exendin-4 Fc fusion protein injection(1.2mg）+Metformin (Experimental): 1.2mg,Subcutaneous injection in the abdomen,Bi-weekly for 54 weeks.
  Interventions: Drug: Exendin-4 Fc fusion protein injection(1.2mg）; Drug: Metformin
- Exendin-4 Fc fusion protein injection(2.4mg）+Metformin (Experimental): The first dose of 1.2 mg of JY09 injection was administered, the dose was adjusted to 2.4 mg after two weeks, after which 2.4 mg was maintained to continue subcutaneous injection in the abdomen, bi-weekly treatment for 52 weeks.
  Interventions: Drug: Exendin-4 Fc fusion protein injection（2.4mg）; Drug: Metformin
- Dulaglutide+Metformin (Active Comparator): 1.5 mg dulaglutide injection subcutaneously once a week for 26 weeks.
  Interventions: Drug: Dulaglutide; Drug: Metformin

INTERVENTIONS:
Drug: Exendin-4 Fc fusion protein injection(1.2mg） — 1.2mg, subcutaneous injection in the abdomen, biweekly, 54 weeks of treatment.
  Other Names: JY09(1.2mg)
  Arms: Exendin-4 Fc fusion protein injection(1.2mg）+Metformin
Drug: Exendin-4 Fc fusion protein injection（2.4mg） — The first dose of 1.2 mg was administered subcutaneously in the abdomen, and after two weeks, the dose was adjusted to 2.4 mg, followed by a continuation of treatment for 52 weeks.
  Other Names: JY09(2.4mg)
  Arms: Exendin-4 Fc fusion protein injection(2.4mg）+Metformin
Drug: Dulaglutide — 1.5 mg dulaglutide injection subcutaneously once a week for 54 weeks.
  Arms: Dulaglutide+Metformin
Drug: Metformin — Metformin hydrochloride tablets, oral administration, 54 weeks of treatment

SUMMARY:
The aim of the study is to compare the efficacy and safety of two JY09 doses versus dulaglutide as add-on therapy to metformin in participants with type 2 diabetes mellitus (T2DM)

DETAILED DESCRIPTION:
This study was designed as a multicenter, randomized, open, parallel, positively controlled Phase III clinical study to evaluate the efficacy and safety of Exendin-4Fc fusion protein (JY09) injection in adult subjects with type 2 diabetes mellitus who have poor glycemic control after metformin treatment only.

The proposed plan is to enroll 600 subjects with T2DM, using stratified block group randomization with the stratification factor being baseline HbA1c (≤8.5% or >8.5%), and randomly assign them to the 1.2 mg JY09 injection group (n=200 subjects), 2.4 mg JY09 injection group (n=200 subjects) and dulaglutide injection group (n=200 subjects) in a 1:1:1 ratio.

The trial was divided into 4 phases, i.e., a screening period of 2 weeks, an introduction period of 4 weeks, a treatment period of 54 weeks (26 weeks for the core treatment period and 28 weeks for the extended treatment period), and a safety follow-up period of 4 weeks. A total of 64 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age and ≤75 years of age at the time of signing the informed consent form.
2. Those who meet the World Health Organization（WHO）1999 diagnostic criteria for type 2 diabetes mellitus and the WHO Recommendations for the Use of Glycosylated Haemoglobin (HbA1c) for Diagnosis (2011) supplemental diagnostic criteria for a diagnosis of T2DM for ≥ 12 weeks.
3. Received a stable dose of metformin monotherapy with a metformin dose ≥1500 mg/day or a maximally tolerated dose (<1500 mg/day but ≥1000 mg/day) on the basis of dietary and exercise interventions during the 8 weeks prior to screening.
4. HbA1c ≥7.5% and ≤11.0% at screening (local laboratory) and HbA1c ≥7.0% and ≤10.5% before randomization (V3) (central laboratory).
5. FPG 13.9 mmol/L at screening (local laboratory) and FPG 13.9 mmol/L before randomization (V3) (central laboratory).
6. Body mass index (BMI) ≥18.5 kg/m2 and ≤35.0 kg/m2 at screening and before randomization (V4).
7. Able to understand and willing to sign a written informed consent form (ICF) and comply with the study protocol.

Exclusion Criteria:

1. People diagnosed with type 1 diabetes or other types of diabetes.
2. Those who have used glucose-lowering drugs other than metformin within 8 weeks prior to screening or prior to randomization (V4), or those who have used drugs that may affect glucose metabolism, such as systemic glucocorticosteroids (except for inhalation or topical topical use) and growth hormone.
3. Those who have used glucose-dependent insulinotropic polypeptide (GIP) and/or glucagon-like peptide-1 (GLP-1) receptor agonists (including single-target, multi-target agonists, and insulin-containing GLP-1 combinations) within 3 months prior to screening.
4. More than 14 days of continuous insulin use in the 6 months prior to screening.
5. Acute complications of diabetes such as diabetic ketoacidosis or hyperglycemic hyperosmolar state within 6 months prior to screening or prior to randomization .
6. Severe chronic complications of diabetes mellitus (e.g., proliferative diabetic retinopathy, severe diabetic neuropathy, diabetic foot, etc.) within 6 months prior to screening, which are assessed by the investigator to be unsuitable for participation in this clinical study.
7. Individuals who have had severe gastrointestinal disease (e.g., active ulcer, gastroparesis, pyloric obstruction, inflammatory bowel disease, etc.) or have undergone gastrointestinal surgery within 6 months prior to screening or prior to randomization or who have been using long-term medications for chronic gastrointestinal disease that have a direct effect on gastrointestinal motility are not suitable for participation in this clinical study, as assessed by the investigator.
8. Other conditions that, in the judgment of the investigator, make the subject unsuitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline, Week 26
  Change in glycated hemoglobin (HbA1c) values relative to baseline after 26 weeks of treatment

SECONDARY OUTCOMES:
The proportion of HbA1c <6.5% and <7% | Baseline, Week 26,Week 54
  Proportion of subjects with HbA1c <7% and HbA1c <6.5% after 26 and 54 weeks of treatment
HbA1c | Baseline, Week 6,Week 10,Week 14,Week 20,Week 38,Week 54
  Change in HbA1c relative to baseline after 6, 10, 14, 20, 38, and 54 weeks of treatment.
fasting plasma glucose (FPG) | Baseline, Week 6,Week 10,Week 14,Week 20,Week 38,Week 54
  Change in fasting plasma glucose (FPG) relative to baseline after 6, 10, 14, 20, 38, and 54 weeks of treatment.
fasting insulin | Baseline, Week 14,Week 26,Week 54
  Change in fasting insulin relative to baseline after 14, 26, and 54 weeks of treatment.
Homeostatic Model Assessment of Insulin Resistance(HOMA-IR) | Baseline,Week 26,Week 54
  Change in HOMA-IR relative to baseline after 26 and 54 weeks of treatment.
Health Survey Short Form (SF-36) | Baseline,Week 26,Week 54
  Value of change in Health Survey Short Form (SF-36) scores relative to baseline after 26 and 54 weeks of treatment.
blood pressure | Baseline,Week 26,Week 54
  Change in blood pressure (sitting) relative to baseline after 26 and 54 weeks of treatment.
  The blood pressure includes systolic and diastolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Junqing Zhang, Doctor, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No